CLINICAL TRIAL: NCT06970002
Title: Assessment of the Importance of Respiratory Stabilization in Patients With Chronic Respiratory Acidosis Before a Diagnostic Bronchofiberoscopy, as Well as the Effectiveness of Different Types of Non-invasive Ventilation During the Procedure
Brief Title: Respiratory Stabilization in Chronic Acidosis Before Bronchofiberoscopy & Non-Invasive Ventilation Effectivenes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BNW/NWN/0052/KB1/95/I/24/25
Record Dates: First submitted 2025-04-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Chronic Respiratory Acidosis
Keywords: Bronchofiberoscopy (FOB); High Flow Nasal Cannula (HNFC); Non-Invasive Ventilation (NIV); Passive Oxygen Therapy; Lung Disease Diagnosis; Chronic Respiratory Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- No respiratory stabilization before FOB: HFNC (Active Comparator): The use of HFNC in pateints with chronic respiratory acidosis undergoing diagnostic FOB without stabilizing their respiratory paramethers before the procedure (pH 7.35-7.45; pCO2 >45 mmHg; HCO3- > 27 mmol/l) HFNC settings: flow 60L/min, temperature 34 ºC and FiO2 under saturation control to achieve SpO2≥ 92%,
  Interventions: Device: Use of HFNC during FOB as a respiratory support method
- No respiratory stabilization before FOB: NIV (Active Comparator): The use of NIV in pateints with chronic respiratory acidosis undergoing diagnostic FOB without stabilizing their respiratory paramethers before the procedure (pH 7.35-7.45; pCO2 >45 mmHg; HCO3- > 27 mmol/l) NIV settings: ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (expiratory positive pressure) 6-12 cmH2O, Tins (duration) 0.8-1.1s, PS 12-23 cm H2O and oxygen flow under saturation control to achieve SpO2≥ 92%
  Interventions: Device: Use of NIV during FOB as a respiratory support method
- Respiratory stabilization before FOB: HFNC (Active Comparator): Use of HFNC during FOB as a respiratory support method The use of HFNC in pateints with chronic respiratory acidosis undergoing diagnostic FOB with stabilization of their respiratory paramethers before the procedure (pH 7.35-7.45; pCO2 35-45 mmHg; HCO3- >27 mmol/l) HFNC settings: flow 60L/min, temperature 34 ºC and FiO2 under saturation control to achieve SpO2≥ 92%,
  Interventions: Device: Use of HFNC during FOB as a respiratory support method
- Respiratory stabilization before FOB: NIV (Active Comparator): The use of NIV in pateints with chronic respiratory acidosis undergoing diagnostic FOB with stabilization of their respiratory paramethers before the procedure (pH 7.35-7.45; pCO2 35-45 mmHg; HCO3- >27 mmol/l) NIV settings: ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (expiratory positive pressure) 6-12 cmH2O, Tins (duration) 0.8-1.1s, PS 12-23 cm H2O and oxygen flow under saturation control to achieve SpO2≥ 92%
  Interventions: Device: Use of NIV during FOB as a respiratory support method
- Respiratory stabilization before FOB: passive oxygen (No Intervention): The use of passive oxygen in pateints with chronic respiratory acidosis undergoing diagnostic FOB with stabilization of their respiratory paramethers before the procedure (pH 7.35-7.45; pCO2 35-45 mmHg; HCO3- >27 mmol/l)

INTERVENTIONS:
Device: Use of NIV during FOB as a respiratory support method — The aim of this project is to assess the safety, indications and contrindications to perform bronchofiberoscopy for diagnostic purposes in patient with chronic respiratory acidosis with the use of Non-invasive Ventilation (NIV) and High Flow Nasal Cannula (HNFC). In addition we want to determine the extent to which the usage of respiratory support during bronchofiberoscopy (BF) will help to avoid complications such as hypoxemia, decompensation of chronic respiratory failure, deterioration of gas exchange and hemodynamic instability, as well as intubation.
  Arms: No respiratory stabilization before FOB: NIV; Respiratory stabilization before FOB: NIV
Device: Use of HFNC during FOB as a respiratory support method — The aim of this project is to assess the safety, indications and contrindications to perform bronchofiberoscopy for diagnostic purposes in patient with chronic respiratory acidosis with the use of Non-invasive Ventilation (NIV) and High Flow Nasal Cannula (HNFC). In addition we want to determine the extent to which the usage of respiratory support during bronchofiberoscopy (BF) will help to avoid complications such as hypoxemia, decompensation of chronic respiratory failure, deterioration of gas exchange and hemodynamic instability, as well as intubation.
  Arms: No respiratory stabilization before FOB: HFNC; Respiratory stabilization before FOB: HFNC

SUMMARY:
Bronchofiberoscopy (FOB) is a minimally invasive and safe procedure performed for diagnostic and therapeutic purposes. FOB frequently impairs respiratory function, which may lead to possible exacerbation of respiratory failure.

Currently, the most frequent respiratory support is passive oxygen therapy, but non-invasive ventilation (NIV) and high flow nasal cannula (HFNC) are increasingly attempted, however the optimal setting and indications for NIV and HFNC in patients undergoing FOB with respiratory acidosis, haven't been determined yet.

Methods:

The study protocol describes a prospective, multicenter, two- armed randomized controlled trial (RCT).

The investigators aim to study two patients groups, based on FOB indications and the type of respiratory acidosis:

1) Diagnostic FOB; patients with chronic respiratory acidosis (pH ≥7.35; pCO2 > 45mmHg and/or HCO3- >27 mmol/l);

1. randomized to: passive oxygen, NIV, HFNC;
2. total number of participants: 210

Randomization:

two-step randomization (1st randomization :a or b; 2nd randomization: i- iii method of respiratory support):

a. Stabilization of respiratory parameters before FOB (pH 7.35-7.45; pCO2 35-45 mmHg; HCO3- >27 mmol/l) i. NIV ii. HFNC iii. Passive oxygen therapy b. FOB right away (pH 7.35-7.45; pCO2 >45 mmHg; HCO3- > 27 mmol/l) i. NIV ii. HFNC

Before FOB, both groups will undergo arterial blood gas analysis (ABG). During FOB there will be a continuous monitoring of vital signs as in: SpO2, FiO2, TcCO2, ECG, and Heart Rate. After FOB, the investigators are going to perform another ABG, mark endpoints, and complications, if any arise.

Results:

Based on the selected endpoints, or any complication related to FOB the investigators hope to determine which of the respiratory methods: passive oxygen, NIV, HFNC or IMV provides the best support, leading to a lower number of complications and overall a better tolerance of FOB by the patient. Additionally, our aim is to find the optimal settings for NIV and HFNC in both studied groups.

Conclusions:

The results of this study are going to assess the need and the role of the optimal respiratory support method among patients with respiratory acidosis, leading to a shorter time from admission to diagnosis, better tolerance during the procedure, quicker recovery after procedure.

DETAILED DESCRIPTION:
Project description Assessment of the importance of respiratory stabilization in patients with chronic respiratory acidosis before undergoing bronchofiberoscopy for diagnostic purposes, as well as the effectiveness of different types of non-invasive ventilation during the procedure.

The aim of the project The aim of this project is to assess the safety, indications and contrindications to perform bronchofiberoscopy for diagnostic purposes in patient with chronic respiratory acidosis with the use of Non-invasive Ventilation (NIV) and High Flow Nasal Cannula (HNFC). In addition the investigators want to determine the extent to which the usage of respiratory support during bronchofiberoscopy (BF) will help to avoid complications such as hypoxemia, decompensation of chronic respiratory failure, deterioration of gas exchange and hemodynamic instability, as well as intubation.

Project justification Bronchofiberoscopy is a minimally invasive procedure performed for diagnostic and therapeutic purposes.

BF is a safe method with high diagnostic value for respiratory diseases. It helps in the diagnosis of hemoptysis, interstitial lung diseases, respiratory system neoplasms and mediastinal lymphadenopathy. In addition, BF can be used therapeutically in cases of foreign body aspiration, airway patency, e.g. in patients with pneumonia or tumors.

BF carries a risk of complications, such as worsening hypoxia, which may contribute to the exacerbation of respiratory failure and secondarily influence the occurrence of cardiac and pulmonary complications.

Sedation improves the patient's tolerance of the procedure, but may contribute to the development of hypoxia and/or respiratory acidosis, which is why various non-invasive mechanical ventilation techniques are more commonly used during the procedure.

The basic method of respiratory support is passive oxygen therapy, although HFNC and NIV are also increasingly used. There are facilities that use HFNC as a standard method of respiratory support. At the moment, there are no clear guidelines published that are supported by experimental data confirming the safety and efficacy of HFNC and NIV in patients with complete respiratory failure who require bronchoscopic procedures.

An important factor for conducting an effective procedure is its good tolerance by the patient, which includes proper blood oxygenation and stable hemodynamic function during the procedure. Inadequate oxygen support ensures the maintenance of proper saturation, whilst the patient may develop acute respiratory acidosis during this time resulting from hypoventilation secondary to the procedure and/or sedation. For this reason, it is important to determine the optimal principles of respiratory support that will allow sedation and BF to be performed with good tolerance and minimizing the risk of complications, because patients with lung diseases such as chronic obstructive pulmonary disease (COPD) or heart failure are particularly susceptible to developing significant hypercapnia during sedation.

NIV is increasingly used to support BF. It prevents atelectasis, reduces the muscle effort associated with breathing, which alleviates dyspnea and the risk of respiratory failure, and also allows for ensuring a normal respiratory rate in a patient undergoing sedation. NIV additionally reduces the risk of serious complications after heart, thoracic and abdominal surgeries. NIV allows for safe performance of diagnostic and therapeutic BF in patients with exacerbation of respiratory failure and in patients with severe chronic respiratory failure.

HFNC is a respiratory support method that allows for obtaining a controlled amount of oxygen in the respiratory mixture - FiO2 with values up to 1.0 (100%). High air flow is associated with other significant advantages of this method - generating a constant, small positive pressure in the airways (CPAP), and washing out respiratory gases from the anatomical dead space, which additionally supports the treatment of total respiratory failure, and functions as air heating and humidification improve the patient's comfort.

NIV and HFNC are used to increase the safety of BF in patients with respiratory failure. This would indicate the possibility of using these methods of respiratory support during diagnostic BF in patients with chronic respiratory acidosis. In patients with acute acidosis or exacerbation of chronic respiratory acidosis, diagnostic BF should be performed after compensation of acidosis.

Currently, there is no evidence to suggest that NIV-BF and/or HFNC-BF are superior in patients with chronic respiratory acidosis. There are also no designated device settings for patients with compensated respiratory acidosis.

Detailed indications and contraindications for performing the above-mentioned procedures have not been determined, nor have the optimal parameters of respiratory support in patients with chronic respiratory acidosis been established.

So far, in this group, intubation has been considered before the procedure in order to safely perform bronchofiberoscopy. Performing BF in an intubated patient results in critical narrowing of the airways, which necessitates mechanical ventilation with the use of high therapeutic pressures, which may result, among others, in barotrauma (injury of the lungs caused by change in air pressure). Because the standard bronchofiberscope fills the lumen of the endotracheal tube almost completely, and the examination can only be performed in patients intubated with a tube of 8 mm or larger in diameter. Small patients, including women, may require intubation with a narrower tube, and in such cases the only solution is to use a pediatric or ultrathin bronchoscope.

In patients who have not been intubated, BF may cause exacerbation of respiratory failure, which may lead to the need for urgent intubation and transfer to the ICU. This complication is extremely rare, as most patients are disqualified from BF.

The possibility of performing BF without the need to equalize blood gas parameters before the procedure may allow for increased access to diagnostics and a reduction in the frequency of intubation of patients.

The study was designed as a multicenter, international prospective randomized controlled trial (RCT). Blood gas analysis will be performed before randomization to confirm chronic respiratory acidosis.

The experiment will be conducted in the respiratory wards participating in the study.

Therefore, the use of NIV and HFNC in patients requiring diagnostic BF who have chronic respiratory acidosis is a research area of potentially great clinical importance.

Silesian Medical University Bioethics Committee (SUM BC) approved the protocole, Resolution No: BNW/NWN/0052/KB1/95/I/24/25

Aim of the study:

* Verification of the role of HFNC, NIV in increasing the safety and availability of bronchoscopic examinations,
* Attempt to determine indications and contraindications to specific respiratory support techniques in patients with indications for BF and chronic respiratory acidosis: HFNC-BF, NIV-BF,
* Attempt to determine the optimal settings for patients with chronic respiratory acidosis undergoing bronchoscopic procedures: HFNC, NIV.

Study group

The study will include patients (women and men) who express informed consent to participate in the proposed study. Recruitment will be conducted in people ≥18 years of age with indications for bronchofiberoscopy for diagnostic purposes.

An interview will be conducted with patients in conditions of privacy and meeting the GDPR criteria. Patients will be thoroughly informed about the course of the study, encouraged to ask questions, with full explanation of doubts. Then, patients will be asked to provide written consent to participate in the research project.

The target planned number of 210 patients studied from all groups (105 patients in each) was calculated based on the risk of complications in the form of intubation during BF in patients with respiratory failure with a frequency estimated at 0.2-2%.

Study population:

COPD, Kyphoscoliosis, Obesity hypoventilation syndrome (OHS), Heart failure, Pulmonary arterial hypertension and the presence of indications for diagnostic BF.

Inclusion criteria:

1. Patient ≥ 18 years of age with indications for diagnostic bronchoscopy:

   ◦ Diagnostic test: suspected lung cancer, suspected sarcoidosis, mediastinal lymphadenopathy,
2. Patient who signed a written informed consent to participate in the study,
3. pCO2 > 45 mmHg and/or HCO3- > 27 mmol/l but pH ≥ 7.35 in a blood gas test performed immediately before qualification for bronchoscopy.

Exclusion criteria

1. Lack of written informed consent of the subject to participate in the research project,
2. Coronary artery disease CCS III/IV,
3. Hemodynamic failure, use of pressor amines, myocardial infarction in the last 2 weeks without PCI treatment, unstable angina pectoris, severe arrhythmias - especially ventricular,
4. Pneumothorax not secured with drainage,
5. Platelet count <20,000/µl, if platelets are not transfused immediately before/during the procedure,
6. INR > 1.5xULN or APTT >36 s.1.5xULN, in the case of diagnostic FOB,
7. Anemia: hemoglobin (Hb) level <6 g/dl or 6-10 g/dl if the physician prescribes a blood transfusion,
8. Patients who were intubated before randomization.

Research methodology A detailed medical history will be collected from the patients (including comorbidities, medications they are taking, smoking history, and NYHA, modified medical research council (mMRC), Charlson's scale, Borg's scale, acute physiology and chronic health evaluation II (Apache II), simplified acute physiology score II (SAPS II), Richmond agitation-sedation scale (RASS) questionnaires). In case of patients undergoing diagnostic FOB a pulmonary function tests (spirometry) will be performed if the patient's clinical condition allows performing it. Blood pressure, saturation, and arterial blood gases (approximately 2.0 ml) will be measured. Arterial blood gases before and after the test. After the patient has been qualified to a specific group, they will be randomly assigned to a given method of respiratory support.

Course of the study and escalation of therapy In the case of high-flow nasal oxygen therapy, the patient will be fitted with special nasal cannulas and then the examination will be performed. In the case of NIV, the patient will be fitted with a non-invasive ventilation mask with a special bronchoscopic elbow containing a valve enabling the introduction of the bronchofiberscope. The examination will compare the initial settings of the devices, which will be maintained provided that the examination is carried out correctly and the patient's clinical condition is stable. In the case of desaturations, hypercapnia or other abnormalities in the assessment of the patient, the settings may be changed or the method may be converted on the basis of therapy escalation (HFNC → NIV).

Monitoring During the entire examination, parameters such as SpO2, FiO2, TcCO2, ECG and heart rate (these parameters will be monitored continuously) as well as arterial blood pressure using a non-invasive method (measured every 5 minutes) will be monitored.

BF will be performed using optical or video bronchofiberscopes or endobronchial endosonography (EBUS) devices. The diameter of the bronchofiberscope used should be noted as well as the type and dose of sedation used during BF in each of the three randomized groups, although bearing in mind that the depth of sedation should be within the RASS range of 0 to -3.

After BF

After the bronchofiberoscopy, arterial blood gasometry will be repeated and the subjects will be assessed at the end of the occurrence of the assumed endpoints.

Data obtained from the interview and additional tests will be anonymously entered into a computer database in accordance with the GDPR criteria and then statistically processed. Appropriate conclusions will be drawn based on the obtained results.

Randomization Randomization will be performed. The database and online randomization platform will be assessable for participating centers online at www.pneumosilesia.org available for collaborating centers after receiving their BC approval.

The patients undergoing a diagnostic FOB there will be a two-step randomization, firstly they will be randomized into two categories deciding if they should be firstly stabilized in terms of respiratory parameters, or not.

Two-step randomization (1st randomization :a or b; 2nd randomization: i- iii method of respiratory support):

a. Stabilization of respiratory parameters before FOB (pH 7.35-7.45; pCO2 35-45 mmHg; HCO3- >27 mmol/l) i. NIV ii. HFNC iii. Passive oxygen therapy b. FOB right away (pH 7.35-7.45; pCO2 >45 mmHg; HCO3- > 27 mmol/l) i. NIV ii. HFNC Device settings

1. HFNC, flow 60L/min, temperature 34 ºC and FiO2 under saturation control to achieve SpO2≥ 92%,
2. NIV will be conducted in ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (expiratory positive pressure) 6-12 cmH2O, Tins (duration) 0.8-1.1s, PS 12-23 cm H2O and oxygen flow under saturation control to achieve SpO2≥ 92%,

Project duration: 3 years

Expected Endpoints

* Possibility of using RASS 0 - -3 sedation (patient comfort) despite signs of hypoventilation,
* Increased safety and comfort of BF in patients with respiratory failure (decrease in the number of procedures in which mild and severe complications occurred),
* Lower probability of exacerbation of acidosis in patients in the NIV group,
* Endpoints and complications such as hospitalization time, bronchospasm, hypoxemia episode, decompensated respiratory acidosis, local bleeding, fever, need to interrupt the procedure, intubation and transfer to the ICU, cardiac arrest, pneumothorax, death will be marked.

Measurable endpoints:

1. Hypoxemia, decrease in saturation >5% for more than 30 seconds,
2. PaO2 before and after BF from blood gas analysis,
3. PaO2/FiO2 before and after BF from blood gas analysis,
4. Hypercapnia measured transcutaneously TcCO2, increase in PaCO2 >10 mm Hg for more than 30 seconds during the examination,
5. PaCO2 before and after BF from blood gas analysis,
6. pH before and after BF from blood gas analysis,
7. Drop in pH below 7.35 after the end of the examination,
8. Duration of hospitalization,
9. Time to diagnosis of the diagnosed disease
10. Time to start targeted treatment (surgery, chemotherapy, X-ray, antibiotic, steroid)
11. Nosocomial infections,
12. New cardiac arrhythmia [>30 s - supraventricular; any ventricular (salvo, bigeminy, etc.),
13. Hypotension, below 90/60 or a drop of more than 30% of the initial value,
14. Duration of HNFC and/or NIV therapy after the procedure,
15. Need for escalation of therapy HFNC-> NIV, NIV-> intubation,
16. Premature termination of the procedure,
17. Need for transfer to the ICU,
18. Complications related to the procedure: fever, bronchospasm, glottis damage, pneumothorax, bleeding,
19. Resuscitation,
20. Periprocedural death,
21. Death - long-term follow-up.

Each complication will be described in 3 time intervals (1-during BF, 2-up to 2h after BF, 3-up to 24h after BF). Long-term prognosis will be assessed based on a telephone conversation with study participants and/or their family members/caregivers after the study recruitment is completed. In the absence of contact, survival will be determined based on Electronic Verification of Beneficiaries' Entitlements.

Funding: The work was supported by the Silesian Medical University (BNW-1-118/N/4/K).

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years of age with indications for diagnostic bronchoscopy:

   ◦ Diagnostic test: suspected lung cancer, suspected sarcoidosis, mediastinal lymphadenopathy,
2. Patient who signed a written informed consent to participate in the study,
3. pCO2 > 45 mmHg and/or HCO3- > 27 mmol/l but pH ≥ 7.35 in a blood gas test performed immediately before qualification for bronchoscopy.

Exclusion Criteria:

1. Lack of written informed consent of the subject to participate in the research project,
2. Coronary artery disease CCS III/IV,
3. Hemodynamic failure, use of pressor amines, myocardial infarction in the last 2 weeks without PCI treatment, unstable angina pectoris, severe arrhythmias - especially ventricular,
4. Pneumothorax not secured with drainage,
5. Platelet count <20,000/µl, if platelets are not transfused immediately before/during the procedure,
6. INR > 1.5xULN or APTT >36 s.1.5xULN, in the case of diagnostic FOB [16],
7. Anemia: hemoglobin (Hb) level <6 g/dl or 6-10 g/dl if the physician prescribes a blood transfu-sion,
8. Patients who were intubated before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
HFNC allows to perform a safe diagnostic FOB in patients with chronic hypercapnia (pCO2>45mmHg; pH 7.35-7.45; HCO3- >27mmol/L) | During the procedure, and after up to the arterial blood gas analysis (1day)
  The investiagors aim to determine if using NIV or HFNC instead of passive oxygen support during the procedure in patients with chronic hypercapnia (pCO2>45mmHg, pH 7.35-7.45, HCO3- >27 mmol/L) results in better respiratory stabiliziation during the procedure without the need to escalate respiratory support therapy during and after the procedure, marking endpoints such as:
  * Hypoxemia, decrease in saturation >5% for more than 30 seconds,
  * PO2 before and after FOB from blood gas analysis,
  * PO2/FiO2 before and after FOB from blood gas analysis,
  * Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study,
  * PCO2 before and after FOB from blood gas analysis,
  * pH before and after FOB from blood gas analysis,
  * Need to extend HNFC therapy after FOB - [time in minutes],
  * Need to escalate HFNC therapy -> NIV, NIV -> intubation,
NIV allows to perform a safe diagnostic FOB in patients with chronic hypercapnia (pCO2>45mmHg; pH 7.35-7.45; HCO3- >27mmol/L) | During the procedure, and after up to the arterial blood gas analysis (1day)
  The investiagors aim to determine if using NIV instead of passive oxygen support during the procedure in patients with chronic hypercapnia (pCO2>45mmHg, pH 7.35-7.45, HCO3- >27 mmol/L) results in better respiratory stabiliziation during the procedure without the need to escalate respiratory support therapy during and after the procedure, marking endpoints such as:
  * Hypoxemia, decrease in saturation >5% for more than 30 seconds,
  * PO2 before and after FOB from blood gas analysis,
  * PO2/FiO2 before and after FOB from blood gas analysis,
  * Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study,
  * PCO2 before and after FOB from blood gas analysis,
  * pH before and after FOB from blood gas analysis,
  * Need to extend NIV therapy after FOB - [time in minutes],
  * Need to escalate NIV therapy -> intubation,
Optimal settings for HFNC in patients with chronic hypercapnia undergoing a diagnostic FOB | During the procedure, and after up to the arterial blood gas analysis (1day)
  Primarily the devices will be set to:
  - HFNC: flow 60L/min, temperature 34 ºC and FiO2 under saturation control to achieve SpO2≥ 92%, During FOB all needed changes in settings for a safe procedures will be marked, if the need for that arises.
  Measurment of parameters for the optimal setting choice:
  Hypoxemia, decrease in saturation >5% for more than 30 seconds, PO2 before and after FOB from blood gas analysis, PO2/FiO2 before and after FOB from blood gas analysis, Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study, PCO2 before and after FOB from blood gas analysis,
  A comaparison of BGA before and after the procedure will allow to determine if those settings and the method itself performs well.
Optimal settings for NIV in patients with chronic hypercapnia undergoing a diagnostic FOB | During the procedure, and after up to the arterial blood gas analysis (1day)
  Primarily the device will be set to:
  NIV will be conducted in ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (expiratory positive pressure) 6-12 cmH2O, Tins (duration) 0.8-1.1s, PS 12-23 cm H2O and oxygen flow under saturation control to achieve SpO2≥ 92%, During FOB all needed changes in settings for a safe procedures will be marked, if the need for that arises.
  Measurment of parameters for the optimal setting choice:
  Hypoxemia, decrease in saturation >5% for more than 30 seconds, PO2 before and after FOB from blood gas analysis, PO2/FiO2 before and after FOB from blood gas analysis, Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study, PCO2 before and after FOB from blood gas analysis,
  A comaparison of BGA before and after the procedure will allow to determine if those settings and the method itself performs well.
The number of complications after a diagnostic FOB in patients with chronic hypercapnia | Through study completion, an average of 1 years
  Endpoints and complications such as prolonged hospitalization, bronchospasm, hypoxemia episode, decompensated respiratory acidosis, local bleeding, fever, need to interrupt the procedure, transfer to the ICU, pneumothorax, death will be marked.

SECONDARY OUTCOMES:
NIV vs HFNC, is one better then the other to support a diagnostic BF in patients with chronic hypercapnia | Through study completion, an average of 1 year
  Secondary outcome, provided the primary outcomes show a good tolerance of both methods is the comparison of respiratory paramethers and analysis of NIV and HFNC, and finding a new standard for the procedure in patients with chronic hypercapnia
  * PO2 before and after FOB from blood gas analysis,
  * PO2/FiO2 before and after FOB from blood gas analysis,
  * Hypoxemia, decrease in saturation >5% for more than 30 seconds
  * Hypercapnia measured transcutaneous TcCO2 during the procedure, increase in PCO2 >10 mm Hg for more than 30 seconds during the procedure,
  * PCO2 before and after FOB from blood gas analysis,
  * pH before and after FOB from blood gas analysis,

CONTACTS AND LOCATIONS:
Overall Officials: Szymon Skoczyński, PhD, professor of university, Principal Investigator — Department of Lung Diseases and Tuberculosis, Faculty of Medical Sciences in Zabrze, Medical University of Silesia, Katowice, Poland.

REFERENCES:
- [Background] Danel A, Tobiczyk E, Warcholinski A, Trzaska-Sobczak M, Swinarew A, Brozek G, Trejnowska E, Batura-Gabryel H, Jedynak A, Scala R, Barczyk A, Cofta S, Skoczynski S. May noninvasive mechanical ventilation and/ or continuous positive airway pressure increase the bronchoalveolar lavage salvage in patients with pulmonary diseases? Randomized clinical trial - Study protocol. Adv Med Sci. 2023 Sep;68(2):482-490. doi: 10.1016/j.advms.2023.10.009. Epub 2023 Nov 7. PMID 37945441
- [Background] Fu ES, Downs JB, Schweiger JW, Miguel RV, Smith RA. Supplemental oxygen impairs detection of hypoventilation by pulse oximetry. Chest. 2004 Nov;126(5):1552-8. doi: 10.1378/chest.126.5.1552. PMID 15539726
- [Background] Skoczynski S, Ogonowski M, Tobiczyk E, Krzyzak D, Brozek G, Wierzbicka A, Trzaska-Sobczak M, Trejnowska E, Studnicka A, Swinarew A, Kucewicz-Czech E, Gierek D, Rychlik W, Barczyk A. Risk factors of complications during noninvasive mechanical ventilation -assisted flexible bronchoscopy. Adv Med Sci. 2021 Sep;66(2):246-253. doi: 10.1016/j.advms.2021.04.001. Epub 2021 Apr 20. PMID 33892212
- [Background] Skoczynski S, Minarowski L, Tobiczyk E, Oraczewska A, Glinka K, Ficek K, Mroz R, Barczyk A. Noninvasive Ventilation-Facilitated Bronchofiberoscopy in Patients with Respiratory Failure. Adv Exp Med Biol. 2019;1160:53-64. doi: 10.1007/5584_2019_375. PMID 30989590
- [Background] Oraczewska A, Cofta S, Warcholinski A, Trejnowska E, Brozek G, Swinarew A, Stolz D, Scala R, Barczyk A, Skoczynski S. The use of non-invasive respiratory assistance to facilitate bronchofiberoscopy performance in patients with hypoxemic (type one) respiratory failure - Study protocol. Adv Med Sci. 2023 Sep;68(2):474-481. doi: 10.1016/j.advms.2023.10.011. Epub 2023 Nov 7. PMID 37945440
- [Background] Qanash S, Hakami OA, Al-Husayni F, Gari AG. Flexible Fiberoptic Bronchoscopy: Indications, Diagnostic Yield and Complications. Cureus. 2020 Oct 24;12(10):e11122. doi: 10.7759/cureus.11122. PMID 33133790